CLINICAL TRIAL: NCT04495647
Title: Feasibility and Safety of Whole-Body Electromyostimulation (WB-EMS) in Frail Older People: A Pilot Study
Brief Title: Feasibility of WB-EMS in Frail Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Paracelsus Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETAPPEN_Pilot
Record Dates: First submitted 2020-07-10; First posted 2020-08-03 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Frailty; Mobility Limitation
MeSH Terms: conditions — Frailty; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: frail older people (n=10) pre-post; robust older (n=10) and young (n=10) reference groups with identical intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WB-EMS_frail (Experimental)
  Interventions: Other: Whole-Body Electromyostimulation
- WB-EMS_robust (Active Comparator)
  Interventions: Other: Whole-Body Electromyostimulation
- WB-EMS_young (Active Comparator)
  Interventions: Other: Whole-Body Electromyostimulation

INTERVENTIONS:
Other: Whole-Body Electromyostimulation — Whole-Body Electromyostimulation (WB-EMS): Simultaneous, individually adjustable stimulation of 12 muscle groups using an interval approach with a duty cycle of 6s impulse/4s rest, bipolar electric current (impulse -frequency 85Hz, -width 350μs, rectangular pattern) will be applied.
  After a 4-week conditioning period, 1.5x 20 min/week WB-EMS will be conducted for 4 weeks (total training duration 8 weeks). Easy to perform functional exercises focusing on balance, transfer ability, stepping and lower extremity strength/power will be done during WB-EMS. Exercise intensity will be individually prescribed and adjusted by rate of perceived exertion (RPE-Borg CR10 scale 4 (moderate) to 7 (hard)).
  WB-EMS will be fully supervised one on one.
  All three arms will receive the same intervention.

SUMMARY:
Exercise in general and resistance training (RT) in particular have demonstrated positive effects on physical functioning and frailty. However, frail older people with functional impairments are among the least physically active and may have problems reaching high intensity levels. The use of special vests with integrated electrodes allows the simultaneous innervation of all large muscle groups by external electrical stimulation, inducing a high-intensity RT at low subjective effort level. This whole-body electromyostimulation (WB-EMS) may be a feasible option inducing training stimuli for functionally impaired frail older people.

This study aims at investigating the feasibility and safety of WB-EMS in frail older people with functional limitations. To explore the effects of age and functional status, young and robust old reference groups will serve as comparators.

ELIGIBILITY:
Frail people

Inclusion Criteria:

* 75+ years
* Frail
* able to walk 4m w/o walking aid
* no prior WB-EMS exposure

Exclusion Criteria:

* severe visual or hearing impairments
* major cognitive impairment (MMSE <10)
* medications with muscle-anabolic effects
* medical conditions affecting trainability of muscles (e.g. Myasthenia gravis, Cushing syndrome, Morbus McArdle)
* surgery within past two months
* history of rhabdomyolysis
* medical conditions affecting sensation of electrical stimuli (e.g. severe polyneuropathy)
* severe renal insufficiency (eGFR<30 ml/min/1.73m²)
* electronic implants
* acute or untreated abdominal wall or inguinal hernia

Robust people

Inclusion Criteria:

* 75+ years
* Robust
* no prior WB-EMS exposure

Exclusion Criteria:

* severe visual or hearing impairments
* major cognitive impairment (MMSE <10)
* medications with muscle-anabolic effects
* medical conditions affecting trainability of muscles (e.g. Myasthenia gravis, Cushing syndrome, Morbus McArdle)
* surgery within past two months
* history of rhabdomyolysis
* medical conditions affecting sensation of electrical stimuli (e.g. severe polyneuropathy)
* severe renal insufficiency (eGFR<30 ml/min/1.73m²)
* electronic implants
* acute or untreated abdominal wall or inguinal hernia

Younger people

Inclusion Criteria:

* 18-50 years
* Healthy
* no prior WB-EMS exposure

Exclusion Criteria:

* severe visual or hearing impairments
* major cognitive impairment (MMSE <10)
* medications with muscle-anabolic effects
* medical conditions affecting trainability of muscles (e.g. Myasthenia gravis, Cushing syndrome, Morbus McArdle)
* surgery within past two months
* history of rhabdomyolysis
* medical conditions affecting sensation of electrical stimuli (e.g. severe polyneuropathy)
* severe renal insufficiency (eGFR<30 ml/min/1.73m²)
* electronic implants
* acute or untreated abdominal wall or inguinal hernia
* pregnancy

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 8 weeks
  measured by ratio of included/eligible participants
Compliance | from baseline to 8 weeks
  measured by proportion of attended training sessions
Retention rate | at 8 weeks
  measured by proportion of participants remaining in the study
Dropout rate | from baseline to 8 weeks
  measured by the proportion of participants not completing the study
Perceived enjoyment measured by the Physical Activity Enjoyment Scale for Older Adults (PACES-8) | Change from baseline to 8 weeks
  The PACES-8 comprises of 8 items on a 7-point bipolar rating scale. A sum score is calculated with higher PACES scores reflecting greater levels of enjoyment.
Intervention engagement measured by the Hopkins Rehabilitation Engagement Scale (HRERS) | at 8 weeks
  The HRERS, reported by instructors, comprises of 5 items on a verbal rating scale from 'Never' to 'Always'. Higher scores reflect greater levels of engagement.
Concentration of Myoglobin (MB) | measured at baseline to week 1, week 3 and week 8
  Concentration of MB measured in µg/l 3 hours after training
Concentration of Creatinkinase (CK) | measured at baseline to week 1, week 3 and week 8
  Concentration of CK measured in U/l before, 48, 72 hours after training
estimated glomerular filtration rate (eGFR) | measured at baseline to week 1, week 3 and week 8
  eGFR (creatinine clearance) measured in mL/min/1.73m² before, 48, 72 hours after training

SECONDARY OUTCOMES:
Rhabdomyolysis surveillance measured by a self-developed questionnaire | measured weekly
  The questionnaire is to be filled out before, immediately after and 24 hours following training and containing information on specific (dark urine, muscle weakness, muscle pain) and unspecific (tachycardia, fever, general malaise, nausea, vomiting) symptoms and other adverse events (e.g. falls)
Pain assessed by the Brief Pain Inventory (BPI-SF) | measured at baseline to week 1, week 3 and week 8
  The BPI-SF comprises of 15 items asking questions on pain location, severity and interference and scored from 0 to 10 with higher scores indicating worse outcomes.
Fatigue assessed by the Brief Fatigue Inventory (BFI) | measured at baseline to week 1, week 3 and week 8
  The BFI comprises of 10 items asking questions on fatigue severity and interference and scored from 0 to 10 with higher scores indicating worse outcomes.
System usability measured by the System Usability Scale (SUS) | once at 8 weeks
  The SUS, reported by instructors, comprises of 10 items on a 5-point Likert scale from 1 ('strongly disagree') to 5 ('strongly agree'). Higher scores reflect greater levels of usability.
Lower extremity functioning measured by the Short Physical Performance Battery (SPPB) | Change from baseline to 9 weeks
  The SPPB comprises of three dimensions, balance (static - standing in 3 positions of increasing difficulty by reducing base of support for max. 10s), gait (usual pace - two walks of 4m lengths), functional strength (chair rise - five times sit-to-stand transfers as fast as possible). A sum score is calculated (0-12 points) with higher scores indicating better functional status and each dimension being equally weighed (0-4 points).
Mobility measured by the Timed up & go test (TUG) | Change from baseline to 9 weeks
  The TUG requires the participants to stand up from chair, walk at usual pace to line at 3m, turn, walk back and sit down again. The time in seconds is recorded.
Maximum knee/hip extension strength | Change from baseline to 9 weeks
  Isokinetic leg press in Newton
Skeletal muscle mass | Change from baseline to 8 weeks
  Bioelectrical impedance analysis (BIA)
Rate of persons with Albuminuria | measured at baseline to week 1, week 3 and week 8
  Rate of persons with Albuminuria ≥ 2+ measured with a semi quantitative urine dipstick 24 hours after training
Rate of persons with Proteinuria | measured at baseline to week 1, week 3 and week 8
  Rate of persons with Proteinuria ≥ 3+ measured with a semi quantitative urine dipstick 24 hours after training
Concentration of Urea | measured at baseline to week 1, week 3 and week 8
  Concentration of Urea measured in mg/dl before, 48, 72 hours after training
Concentration of Cystatin C | measured at baseline to week 1, week 3 and week 8
  Concentration of Cystatin C measured in mg/l before, 48, 72 hours after training
Concentration of Creatinine | measured at baseline to week 1, week 3 and week 8
  Concentration of Creatinine measured in mg/dl before, 48, 72 hours after training
Concentration of Sodium | measured at baseline to week 1, week 3 and week 8
  Concentration of Sodium measured in mmol/l before, 48, 72 hours after training
Concentration of Potassium | measured at baseline to week 1, week 3 and week 8
  Concentration of Potassium measured in mmol/l before, 48, 72 hours after training
Concentration of Calcium | measured at baseline to week 1, week 3 and week 8
  Concentration of Calcium measured in mmol/l before, 48, 72 hours after training
Concentration of Phosphate | measured at baseline to week 1, week 3 and week 8
  Concentration of Phosphate measured in mmol/l before, 48, 72 hours after training

OTHER OUTCOMES:
Health-related quality of life measured by the patient-reported Health Survey Short Form (SF-12) | Change from baseline to 9 weeks
  The SF-12 comprises of 12 items weighted and summed to provide physical and mental health scores (PCS and MCS), ranging from 0 to 100 with higher scores reflecting greater levels of the respective construct.
Concentration of Interleukin 6 (IL-6) | measured at baseline to week 1, week 3 and week 8
  Concentration of IL-6 measured in ng/l before, 3h, 48, 72 hours after training
Concentration of High-sensitivity C-reactive protein (hs CRP) | measured at baseline to week 1, week 3 and week 8
  Concentration of hs CRP measured in mg/l before, 48, 72 hours after training
Concentration of Cholesterin | measured at baseline and week 8
  Concentration of Cholesterin measured in mg/dl before first and last trainings
Concentration of low-density lipoprotein (LDL) | measured at baseline and week 8
  Concentration of LDL measured in mg/dl before first and last trainings
Concentration of high-density lipoprotein (HDL) | measured at baseline and week 8
  Concentration of HDL measured in mg/dl before first and last trainings
Concentration of Triglycerides | measured at baseline and week 8
  Concentration of Triglycerides measured in mg/dl before first and last trainings
Concentration of N-terminal pro b-type natriuretic peptide (NT-proBNP) | measured at baseline to week 1, week 3 and week 8
  Concentration of NT-proBNP measured in pg/ml before, 48, 72 hours after training
Concentration of Glucose | measured at baseline and week 8
  Concentration of Glucose measured in mg/dl before first and last trainings
Concentration of Creatinkinase Muscle/Brain (CK-MB (CK-2)) | measured at baseline to week 1, week 3 and week 8
  Concentration of CK-MB (CK-2) measured in ng/ml before, 48, 72 hours after training
Concentration of high-sensitive cardiac troponin T (hs-cTnT) | measured at baseline to week 1, week 3 and week 8
  Concentration of hs-cTnT measured in ng/ml before, 48, 72 hours after training

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Medical Physics, University of Erlangen-Nürnberg, Erlangen, Germany